CLINICAL TRIAL: NCT04827719
Title: Phase 2, Open-Label, Single Arm, Multi-Center Study to Assess the Efficacy and Safety of BST-236 as a Single Agent in Adults Unfit for Intensive Chemotherapy With Relapsed or Refractory Acute Myeloid Leukemia or HR-MDS .
Brief Title: BST-236 as a Single Agent in Adults With Relapsed or Refractory AML or HR-MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-BST003
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BST-236 (Experimental): Recurrent 6 days treatment courses with BST-236 (4.5 g/m2/d administered IV over 1 hour for 6 consecutive days)
  Interventions: Drug: BST-236

INTERVENTIONS:
Drug: BST-236 — Recurrent 6 days treatment courses with BST-236 (4.5 g/m2/d administered IV over 1 hour for 6 consecutive days)

SUMMARY:
To assess the efficacy, and safety of BST-236 in patients unfit for intensive chemotherapy with AML or HR MDS that failed or relapsed following first line therapy

DETAILED DESCRIPTION:
This is a prospective, phase 2, open-label, multi-center, single arm, single agent study, in unfit adult patients with AML or HR MDS who failed or relapsed following first-line therapy.

The study consists of three periods:

Screening: Up to 28 days Treatment: Recurrent 6 days treatment courses with BST-236 Follow-up: The period of time from last day of BST-236 treatment to completion of one year (365 days ±7 days) from the first day of BST-236 treatment

Post-study Follow-up: The period of time from last day of BST-236 treatment to completion of one year (365 days ±7 days) from the first day of BST-236 treatment

Follow-up: One-Year follow-up of survival, starting at the end of study visit

Treatment period: After signing the Informed Consent Form (ICF), meeting all eligibility criteria, and undergoing screening assessments for up to four weeks, eligible patients will receive the first induction course with BST-236, 4.5 g/m2/d administered IV over 1 hour for 6 consecutive days. The first day of the induction is defined as Study Day 1. Following the first treatment course:

1. AML patients in complete remission (CR) or CR with incomplete count recovery (CRi) or CR with partial hematologic recovery (CRh), and HR MDS patients with CR will receive between 2 to 4 maintenance courses of 6-day treatment with BST-236, every 4-6 weeks. The BST-236 dose in these subsequent treatment courses will be 2.3g /m2/d or 4.5 g/m2/d. The reduced dose must be used in case of previous courses toxicity and is allowed in certain cases according to physician discretion following consultation with the study medical monitor. The interval between treatment courses may be extended to up to 12 weeks to allow resolution of toxicities per investigator discretion and in consultation with principal investigators.
2. Patients with stable disease defined as failure to achieve at least PR, but with no evidence of disease progression or patients in partial response (PR) will receive a second 6-day course with BST-236, at a dose of 4.5 g/m2/d. Following which:

   1. AML patients in PR or CR, (including CR, CRh or CRi) and HR MDS patients in PR or CR will be treated with maintenance courses as detailed above Patients in stable disease or disease progression may receive alternative treatment outside of the protocol and will be followed for overall survival (OS) until the completion of 1 year of participation in the study (365 days±7 days from the first day of BST-236 treatment). Additional 1 year of post study follow-up will be implemented for these patients in order to follow up on their survival status and their current AML/MDS treatments.

Patients that have a disease progression while treated in the maintenance courses, will not receive any additional BST-236 treatment and will be followed until the completion of 1 year of participation in the study. These patients may also receive alternative treatment outside of the protocol, in such case, they will be followed in regular intervals for progression free survival, OS and development of new malignancies.

Follow-up period: All patients will be followed by periodic in person in-clinic visits, until the completion of 1 year of participation in the study (365 days±7 days from the first BST-236 treatment day).

End of Study (EOS) visits: will be performed on the last day of participation in the study for all patients.

Scheduled in-clinic visits to assess safety and efficacy outcomes will be conducted during the study periods as specified in the Schedule of Activities.

Unscheduled visits may be conducted at any time for safety reasons or for any other reason.

Post study follow-up: All patients will be followed for survival for an additional 1 year from the EOS

QT Evaluation with Pharmacokinetics (PK) sub-study: Up to 20 patients participating in the main study in pre-selected sites, will be asked to participate in a QT evaluation with PK sub-study to assess the effect of BST-236 on the cardiac electrophysiology. In this study, up to 14 blood samples for PK analysis will be taken from each patient during the first induction course and a continuous electrocardiogram (ECG) recording by a Holter monitor will be done in the first 24 hours of BST-236 administration. Patients participating in this study will be asked to sign an additional ICF for the collection of the PK blood samples and ECG recording.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Documented diagnosis of MDS, according to World Health Organization (WHO) classification (Appendix 1) and assessed as higher risk MDS, prior to first line hypomethylating agents (HMA) treatment, according to the Revised International Prognostic Scoring System (IPSS-R) (IPSS-R overall score ≥ 4.5) Or Diagnosed AML according to the 2016 revision to the WHO classification of myeloid neoplasms and acute leukemia: ≥20% blasts in peripheral blood or bone marrow
2. Adult ≥18 years of age
3. Failure/relapse following prior first-line AML or MDS treatment, defined as:

   1. For MDS:

      * Relapse after initial complete or partial response or stable disease with hematologic improvement (HI), according to International Working Group (IWG) 2006 criteria following treatment with azacitidine or decitabine Or
      * Failure to achieve complete or partial response or stable disease with hematologic improvement (HI) according to International Working Group (IWG) 2006 criteria after at least 4 cycles of azacitidine or decitabine, all within the last 1 year Or iii. MDS progression while on azacitidine or decitabine treatment irrespective of the number of cycles the patient has received
   2. For AML:

      * Relapse after initial CR/CRi/CRh following treatment with: azacitidine, decitabine, Low-Dose Ara-C (cytarabine) [LDAC] (20 mg/m2/d), venetoclax+HMA, or venetoclax+LDAC Or
      * Failure to achieve CR, CRh or CRi following at least 4 cycles of azacitidine or decitabine or 2 cycles of venetoclax+HMA or venetoclax+LDAC within the last 1 year.

   Or

   - AML progression while on azacitidine, decitabine, LDAC, venetoclax+HMA, venetoclax+LDAC, irrespective of the number of cycles the patient has received.
4. The participant is not able to receive an allogeneic bone marrow transplantation (BMT) at the time of study enrolment (BMT may be an option once the patient completed the study).
5. Not eligible for intensive chemotherapy;

   1. Age ≥75 years Or
   2. Age ≥18 years with at least one of the following comorbidities:

   I. Significant heart or lung comorbidities, as reflected by at least one of the following:
   * Left ventricular ejection fraction (LVEF) ≤50%
   * Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected
   * Forced expiratory volume in 1 second (FEV1) ≤65% of expected II. Other comorbidity that the Investigator judges as incompatible with intensive chemotherapy, which must be documented
6. Creatinine clearance (estimated by the Modification of Diet in Renal Disease (MDRD) equation or measured by 24 hours urine collection) ≥45 mL/min
7. Liver enzymes (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 times the upper limits of normal (ULN), unless attributed to leukemia (in AML patients)
8. Total bilirubin ≤3 XULN unless due to Gilbert disease
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
10. Women of reproductive potential must have a negative serum pregnancy test within 48 hours prior to the first day of any BST-236 treatment course
11. Women of reproductive potential must use two forms of effective birth control methods starting from at least 1 month prior to BST-236 first dose and until 6 months following the last BST-236 administration day (acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, intrauterine hormone-releasing system, long-acting injectable contraceptives, or vasectomized partner (provided that partner is the sole sexual partner)
12. Male subjects must agree to refrain from unprotected sex unless vasectomized and from sperm donation from initial study drug administration until 6 months following the last dose of study drug
13. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures
14. Patient must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

Patients with any one of the exclusion criteria listed below are not eligible for the study:

1. MDS or AML evolving from a pre-existing myeloproliferative neoplasm (MPN)
2. MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN
3. Acute promyelocytic leukemia
4. Previous treatment for AML or MDS with drugs other than HMA or LDAC or combinations of venetoclax with either HMA or LDAC
5. Previous allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation
6. Participation in a previous clinical trial involving use of an investigational drug within 30 days or at least 5 half-lives of tested drug (whichever is shorter) of study day 1
7. Peripheral White Blood Cell (WBC) count >30,000/L in the 48 hours prior to first BST-236 dose administration. Hydroxyurea administration or leukapheresis is permitted to meet this criterion
8. Administration of HMA, LDAC, or venetoclax within 14 days prior to Study Day 1
9. Previous treatment with cytarabine at a dose higher than 20 mg/ m2/d
10. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment)
11. Any medical or surgical condition, presence of laboratory abnormalities or psychiatric illness that may preclude safe and complete study participation based on the Investigator's judgment
12. Diagnosis of malignant disease (other than AML) within the previous 12 months (excluding basal cell carcinoma of the skin without complications, "in-situ" carcinoma, or other local malignancy excised or irradiated with a high probability of cure and not treated with systemic or topical chemotherapy)
13. Surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) in the 14 days prior to first BST-236 dose administration
14. History of allergic reactions attributed to compounds of similar chemical composition as BST-236 and/or cytarabine
15. Life expectancy shorter than 3 months attributed to any known medical condition other than AML/MDS
16. Known infection with Hepatitis B Virus (HBV) Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
17. In 12 leads ECG, corrected QT interval (QTc)>480msec or history of QT prolongation or Torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Overall hematological response | 2 months
  Overall response rate

SECONDARY OUTCOMES:
response duration | 12 months
  response duration

CONTACTS AND LOCATIONS:
Overall Officials: Marie Anne HOSPITAL, MD, Principal Investigator — Institut Paoli Calmettes, Marseille; PIERRE FENAUX, Pr, Principal Investigator — Hôpital St Louis-Paris
Locations (17):
- France (17):
  - CHU NIMES Caremeau, Nîmes, Nîmes
  - Centre Henri Becquerel, Rouen, Rouen
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux Haut-Lévèque, Bordeaux
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - CHRU de Limoges - Hôpital Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital Archet 1, Nice
  - Hôpital Saint Louis, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU Toulouse - IUCT Oncopole, Toulouse